CLINICAL TRIAL: NCT03283007
Title: A Multi-center, Randomised, Double-blind Trial of Nintedanib in Lung Transplant (LTx) Recipients With Bronchiolitis Obliterans Syndrome (BOS) Grade 0p-1-2
Brief Title: Nintedanib in Lung Transplant Recipients With Bronchiolitis Obliterans Syndrome Grade 0p-1-2
Acronym: INFINITx BOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P160907
Record Dates: First submitted 2017-09-06; First posted 2017-09-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: Lung-transplant Recipients
Keywords: Nintedanib, lung transplantation, bronchiolitis obliterans syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nintedanib (Experimental): Eligible LTx recipients with BOS receive Nintedanib treatment at a dose of 150 mg twice daily (bid) for 6 months
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): Eligible LTx recipients with BOS receive Nintedanib 150 mg BID matching placebo treatment for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — Eligible LTx recipients with BOS receive Nintedanib treatment at a dose of 150 mg twice daily (bid) for 6 months
  Arms: Nintedanib
Drug: Placebo — Eligible LTx recipients with BOS receive Nintedanib 150 mg BID matching placebo treatment for 6 months
  Arms: Placebo

SUMMARY:
Lung transplantation (TxP) is now a validated treatment of end-stage pulmonary diseases, but long-term graft and patient survival are still hampered by the development of chronic allograft dysfunction (CLAD) affecting > 50% of patients.

The investigators propose to conduct a phase III clinical randomized trial that will assess the efficacy of Nintedanib to hamper the lung decline in LTx recipients with BOS. This is the first trial testing this molecule in lung Tx recipients. If case of demonstrated effectiveness of Nintedanib, the benefit for lung transplant patients carrying a BO is high in terms of stabilization of lung function and enhancement of survival.

DETAILED DESCRIPTION:
Introduction: Lung transplantation (TxP) is now a validated treatment of end-stage pulmonary diseases, but long-term graft and patient survival are still hampered by the development of chronic allograft dysfunction (CLAD) affecting > 50% of patients. Obliterative bronchiolitis (OB), the obstructive CLAD, is the most common manifestation of CLAD, and affects > 50% of recipients who survive the early post-transplant period. OB is thought to arise from repeated injury to graft epithelial cells, leading to fibrous scarring and obliteration of the small airway lumen, as a result of dysregulated fibrotic repair and loss of peribronchial microvasculature. The patchy histopathologic distribution at onset makes it difficult to confirm histopathologically the diagnosis of OB from lung specimens. Hence, bronchiolitis obliterans syndrome (BOS) has become a generally accepted surrogate diagnostic of OB, characterized physiologically by progressive airflow limitation, with a median monthly decline of FEV1 of about 50 ml. Survival after onset of BOS is poor, reported as < 50% at 3 years after onset of disease, due to end-stage respiratory failure. Thus far, there is currently no approved treatment to stabilize BOS disease, and especially no treatment addressing the fibrotic lung graft manifestation of BOS. The crucial role of a dysregulated fibrotic repair has now been demonstrated in BOS, with the following: (i) Architectural remodelling with fibrosis and scarring of airways involving myofibroblasts; (ii) Increased extracellular matrix synthetic; (iii) Epithelial-mesenchymal transition mechanism; (iv) Role of growth factors PDGF, VEGF, FGF, and IGF-1 shown in BO mechanisms (animals and humans studies).

These data strongly suggest the potential role of tyrosine kinase inhibitors (TKI) that target these growth factors involved in the post-TxP BO. In this axis, the new TKI Nintedanib, which has recently been demonstrated as effective in the treatment of idiopathic pulmonary fibrosis (IPF) in large-scale randomized studies (8) appears as a candidate molecule capable of stopping the fibroproliferative process and stabilize the development of a CLAD after TxP. Whereas Nintedanib is a validated and available treatment in patients with IPF, paucity of data are currently available in lung-transplant recipients.

Primary objective: to assess Nintedanib efficacy in the reduction of the rate of decline of FEV1 (forced expiratory volume in 1 sec) in BOS post-LTx at a dose of 150 mg twice daily (bid) compared to placebo over 6 months.

Secondary objectives: to assess Nintedanib efficacy and tolerance in the treatment of BOS grade 0p-1-2 post-lung transplantation.

Experimental design: a 2 groups parallel, randomized, prospective multicentric placebo-controlled phase III trial to assess Nintedanib superiority versus placebo.

Eligible LTx recipients with BOS are to be randomized in a 1:1 ratio to receive either Nintedanib 150 mg BID or the matching placebo treatment for 6 months.

The follow-up of patients with BOS included in the trial will be similar to usual and standard care in both arms of the study (Nintedanib group and placebo group).

The intervention group is expected to be beneficial compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed prior to entry into the trial
2. Patients ≥18 years of age when signing his/her informed consent
3. Patients at least at 6 months post-LTx
4. Single- or double-LTx or combined cardio-pulmonary LTx are eligible
5. Patients must have diagnosis of BOS defined as a decrement of 10% or more in forced expiratory volume in 1 seconde (FEV1) compared to post-transplant baseline FEV1 individualized for each patient according to ISHLT definition. The documented post-LTx baseline value of FEV1 is defined as the mean of the 2 highest values measured at least 3 weeks apart according to ISHLT criteria, and post-LTx VC measurements
6. Patients must have BOS grade 0p, 1 or 2
7. Patients must have documented progressive BOS as demonstrated by the following criteria: at least 3 FEV1 and VC measurements in the last 12 months prior V1, each at least 3 weeks apart, with a total decline of at least 200ml in FEV1 in these last 12 months AND FEV1/VC<0.7
8. Azithromycin therapy for at least 4 weeks prior to V1, with an Azithromycin dose of minimum 250 mg/day at least 3 times per week as this is considered standard therapy for bronchiolitis obliterans syndrome

Exclusion Criteria:

Related to LTx

1. Criteria of restrictive allograft syndrome (RAS) at V0, including the following: (1) Decline of VC < 20% of best post-LTx value (FVCBest is defined as the average of the two FVCs associated with the two PFTs used in FEV1 baseline calculation for CLAD diagnosis) AND FEV1/VC > 0.7 AND (2) Thorax HRCT at entry demonstrate new significant findings which are compatible with RAS like interstitial fibrosis, consolidation, appearances suggesting Restrictive Allograft Syndrome (RAS)
2. FEV1 and/or FV and/or TLC decline related to other nonCLAD causes (eg Diaphragm dysfunction, pneumothorax or pleural effusion, evolutive bronchial stricture within the previous 3 months)
3. At V0, patients who already have developed severe BOS grade 3
4. Patients with severe comorbidity complicating CLAD which might determine the prognosis and functional level of the patient (e.g. evolutive invasive aspergillosis or mycobacterial infection within the last 3 months, active malignant disease within the last 12 months)
5. At visit V1 (end of screening period), diagnosis of documented acute cellular (AR) perivascular rejection higher than grade A1 within the 4 prior weeks OR diagnosis of acute antibody-mediated rejection within the 4 prior weeks, based on presence of all 4 following criteria: 1) acute lung allograft dysfunction, 2) detection of donor-specific antibodies, 3) histological findings compatible with AMR on transbronchial lung biopsy TBBx, and 4) detection of C4d > 50% on TBBx
6. At visit V1 (end of screening period), diagnosis of documented acute pulmonary infection within the 2 prior weeks, on the basis of the following: 1) clinical, radiological and physiological deterioration; AND 2) isolation of an organism from a clinically relevant BAL fluid culture; AND 3) antibiotic therapy resulting in a full recovery and return to pre-morbid lung function
7. Previous treatment with Nintedanib after the date of lung transplantation (Treatment with Nintedanib before lung transplantation is not an exclusion criteria)
8. Ongoing treatment with photopheresis at V1 or planned treatment with photopheresis within the study period.

   Laboratory parameter thresholds
9. Within the 2 weeks prior to V1, renal insufficiency with following criteria: Creatinine clearance <30 ml/min estimated by the Cockcroft-Gault equation
10. Within the 2 weeks prior to V1, any of the following liver test criteria above the specified limit: Total bilirubin > 1.5 above the upper limit of the normal range (ULN), except in patients with predominantly unconjugated hyperbilirubinemia (e.g., Gilbert's syndrome). Aspartate or alanine aminotransferase (AST or ALT) >3 × ULN (refer to the protocole, for the management of liver enzyme elevation).

    General exclusion criteria
11. Pregnancy or lactation (women of childbearing capacity are required to have a negative serum pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using at least two methods of birth control from the date of consent to three months after the end of the patient study participation)
12. Other investigational therapy received within 1 month or 6 half-lives (whichever was greater) prior to screening visit (V0)
13. Alcohol or drug abuse which in the opinion of the treating physician would interfere with treatment
14. Patients not able to understand and follow study procedures including completion of self-administered questionnaires without help.

    Other diseases
15. Cardiac disease: (1) History of myocardial infarction within 6 months of visit 1 or unstable angina within 6 months of visit 1; (2) Presence of aortic stenosis (AS) per investigator judgement at visit 1; (3) Severe chronic heart failure: defined by left ventricular ejection fraction (EF) < 25% per investigator judgement at visit 1
16. Known allergy or hypersensitivity to Nintedanib or intolerance to nintedanib, peanut or soya, or any other components of the study medication
17. Bleeding Risk: Known genetic predisposition to bleeding; Patients who require fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors, heparin, hirudin, etc.) or high dose antiplatelet therapy (acetyl salicylic acid >325 mg/day, or clopidogrel >75 mg/day) [NB: Prophylactic low dose heparin or heparin flush as needed for maintenance of an indwelling intravenous device (e.g. enoxaparin 4000 I.U. s.c. per day), as well as prophylactic use of antiplatelet therapy (e.g. acetyl salicylic acid up to 325 mg/day, or clopidogrel at 75 mg/day, or equivalent doses of other antiplatelet therapy) are not prohibited]; History of haemorrhagic central nervous system (CNS) event within 12 months prior to visit 1; History of haemoptysis or haematuria within 3 months prior to visit 1, active gastro-intestinal bleeding or ulcers and/or major injury or surgery within 3 months prior to visit 1; International normalised ratio (INR) > 2 at visit 1; Prothrombin time (PT) and activated partial thromboplastin time (aPTT) > 150% of institutional ULN at visit 1
18. Patients with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment)
19. Planned major surgery during the trial participation
20. History of thrombotic event (including stroke and transient ischemic attack) within 6 months of visit 1
21. Second-degree or third-degree atrioventricular (AV) block on electrocardiogram (ECG) per investigator judgement at visit 1
22. i) Hypotension (systolic blood pressure [SBP] < 90 mm Hg or diastolic blood pressure [DBP] < 50 mm Hg) (symptomatic orthostatic hypotension) at visit 1 ii) Uncontrolled systemic hypertension (SBP > 160 mmHg; DBP > 100 mmHg) at visit 1
23. Known penile deformities or conditions (e.g., sickle cell anemia, multiple myeloma, leukemia) that may predispose to priapism
24. Retinitis pigmentosa, or History of vision loss, or History of nonarteritic ischemic optic neuropathy
25. Ongoing treatment with pirfenidone at V1 or planned treatment with pirfenidone within the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Nintedanib efficacy in the reduction of the rate of decline of FEV1 (forced expiratory volume in 1 sec) in BOS post-LTx grade 0p-1-2 at a dose of 150 mg twice daily (bid) compared to placebo over 6 months | 6 months
  The absolute difference of FEV1 in mL over 6 months of treatment defined by the rate of decline between inclusion (Visit 1) and month 6 (Visit 4) will be compared between Nintedanib versus Placebo groups

SECONDARY OUTCOMES:
Nintedanib efficacy on exercise tolerance in LTx recipients | 6 months
  Nintedanib efficacy on exercise tolerance will be assessed by the absolute change from baseline in the 6-min Walking Test at month 6 in Nintedanib group compared to Placebo group
Nintedanib efficacy on quality of life improvement in LTx recipients | 6 months
  Nintedanib efficacy on quality of life improvement will be assessed by the absolute change from baseline in SGRQ (Saint George's Respiratory Questionnaire) total score at month 6 in Nintedanib group compared to Placebo group
Nintedanib efficacy to hamper FEV1 decrease in LTx recipients | 6 months
  Nintedanib efficacy to hamper FEV1 decrease will be assessed by the absolute change of FEV1 in mL at month 6 by a repeated FEV1 measurements (at month 0, month 1, month 3, month 6) in Nintedanib group compared to Placebo group
Nintedanib efficacy to hamper progression of BOS in LTx recipients | 6 months
  Nintedanib efficacity to hamper progression of BOS will be assessed by the proportion of patients with change in BOS grade and graft failure (defined as death or retransplantation) in Nintedanib group compared to Placebo group
Nintedanib efficacy on the change of Oxygen saturation in LTx recipients | 6 months
  Nintedanib efficacity on the change of Oxygen saturation will be assessed by the absolute change from baseline in Oxygen saturation (expressed in percent) rest evaluated from baseline at month 6 in Nintedanib group compared to Placebo group
Nintedanib tolerance in LTx recipients | 6 months
  Nintedanib tolerance in lung-transplant recipients over 6 months will be assessed in comparing occurrence of adverse events between both arms (Nintedanib vs Placebo)
Explanatory parameters of fibrotic pathways | 6 months
  Explanatory parameters of fibrotic pathways will be assessed by absolute changes of biomarkers of alveolar cells injury (Krebs von den Lungen-6 (KL6), surfactant apoprotein D (SPD), and growth factors as vascular endothelial growth factor (VEGF) and platelet-derived growth factor (PDGF)) since baseline at month 6

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Brugière, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Foch Hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: Undecided